CLINICAL TRIAL: NCT02412280
Title: Validity of Different Prognostic Models Assessing 1 Year Survival After Liver Transplantation
Acronym: ProgModels
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, Dr, Mansoura University
Other Study IDs: 6
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: retrospecive observational

SUMMARY:
Validity of MELD vs MELD XI in assessing 1 year survival after living donor liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* liver transplantation recipients

Exclusion Criteria:

* Patient refusal

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: liver failure
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
1 year survival | 1 year